CLINICAL TRIAL: NCT06400355
Title: Effect of Mannitol on Recovery Pattern After Orthognathic Surgery, a Prospective Randomized Double Blind Controlled Study.
Brief Title: Effect of Mannitol on Recovery Pattern After Orthognathic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Collaborators: faculty of medicine, Benha university (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC1-3-2024
Record Dates: First submitted 2024-04-21; First posted 2024-05-06 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Orthognathic Surgery
Keywords: Mannitol; Recovery; Orthognathic Surgery; mandiblular fracture; maxillary protrusion
MeSH Terms: interventions — Mannitol; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: The aim of this study is to test, whether mannitol infusion in will affect recovery pattern?
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which will include 30 patients. Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): in which mannitol will be given in doses of 0.5 gm/kg 30 minutes before the end of the surgery.
  Interventions: Drug: Mannitol
- Group C (Active Comparator): similar volume of the infused mannitol but of lactated Ringer will be given 30 minutes before the end of the surgery
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Mannitol — in which mannitol will be given in doses of 0.5 gm/kg 30 minutes before the end of the surgery
  Arms: Group M
Drug: Ringer's Lactate — similar volume of the infused mannitol but of lactated Ringer will be given 30 minutes before the end of the surgery.
  Arms: Group C

SUMMARY:
The aim of this study is to test, whether mannitol infusion in different doses will affect recovery pattern? the investigators hypothesized that infusion of mannitol in doses of 0.5 gm/kg before recovery from anesthesia after orthognathic surgery shortens patients' recovery time, and improves recovery quality, as well as postoperative cognitive function better.

DETAILED DESCRIPTION:
The aim of this study is to test, whether mannitol infusion in different doses will affect recovery pattern? the investigators hypothesized that infusion of mannitol in doses of 0.5 gm/kg before recovery from anesthesia after orthognathic surgery shortens patients' recovery time, and improves recovery quality, as well as postoperative cognitive function better Methodology This prospective randomized double blinded study will be applied on patients scheduled for orthognathic surgeries as Temporo-mandibular joint procedures, Le Forte Ι 0r II osteotomy, bimax or maxillectomy after ethical committee approval.

The selected patients were randomly allocated into two groups each containing 30 patients:

* Group M: in which mannitol will be given in doses of 0.5 gm/kg 30 minutes before the end of the surgery
* Group C: similar volume of the infused mannitol but of lactated Ringer will be given 30 minutes before the end of the surgery

Anaesthetic technique:

For all Patients, atropine sulphate 0.015 mg/kg intramuscular (IM) as anti-sialgogue together with dexamethasone 8 mg. Hydrocortisone 100 mg and ranitidine 50 mg, will be given IV as pre-medications 15-30 minutes before induction of anaesthesia patient will be transferred to the operating theatre where ASA-basic monitors will be applied to the patient (pulse-oxymitery, non-invasive blood pressure, ECG 3-Leads and capnography).

Induction of anesthesia:

Regular IV induction will be applied for patients with normal mouth opening where difficult intubation is not suspected: fentanyl 2 μg/kg IV, propofol 1 mg/kg IV, atracurium 0.5 mg/kg IV then nasotracheal intubation with armored tube of appropriate size.

Patients with difficult mouth opening will undergo awake fiberoptic intubation. Anesthesia will be maintained by 100% O2 + 1-1.5 MAC isoflurane Thirty minutes before the end of surgery patients will receive an IV solution which is either mannitol 0.5 gm/kg or lactated Ringer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* ASA status I and II patient.
* No contraindication to use of mannitol.

Exclusion Criteria:

* ASA III and IV status
* Extreme of age: paediatric and geriatric patients
* Severe cardio respiratory, rheumatological or endocrinal disorders
* Pregnancy and lactation
* Contraindications to the use of mannitol, e.g. serum osmolality > 330, renal failure systemic hypertension, proved intra-cranial brain haemorrhage or sub-dural haematoma and hypotension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to extubation | 1st 2 hour post-surgery
  Time to extubation which is defined as time from cessation of inhalation anesthetic to extubation

SECONDARY OUTCOMES:
Quality of Recovery-15 (QoR-15) | 1st 2 hour postoperative
  A patient-reported outcome measure measuring quality of recovery after surgery and anaesthesia. It is a 15-point questionnaire with an 11-point numerical rating scale (for positive items, 0 = "none of the time" to 10 = "all of the time"; for negative items the scoring was reversed; maximum score 150).
Time between anesthesia termination and discharge from PACU | 1st hour 2hours postoperative
  Time between anesthesia termination and discharge from PACU
Urine output | 24 hours postoperative
  Urine output

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Soliman, Principal Investigator — National Cancer Institute Cairo university; Mahmoud M kaml, Principal Investigator — National Cancer Institute Cairo university
Locations (1):
- Benha Univesity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till publication